CLINICAL TRIAL: NCT06068569
Title: Safety, Reactogenicity and Immunogenicity Study of the Vector Vaccine GamCovidVac for the Prevention of Coronavirus (COVID-19) Infection Caused by the SARS-CoV-2 Virus With Altered Antigenic Profile With Participation of Adult Volunteers
Brief Title: Study of the Vector Vaccine GamCovidVac for the Prevention of COVID-19 With Altered Antigenic Profile With Participation of Adult Volunteers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12-GamCovidVac/N-2023
Record Dates: First submitted 2023-09-26; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy patients (Experimental): Drug: GamCovidVac vector vaccine for the prevention of COVID-19 (with altered antigenic profile); A total of 50 people will be randomized and receive the study drug (vaccine). Two intramuscular injections of the investigational medicinal product (IMP) will be performed. 1st injection - component I, 2nd injection - component II.
  Interventions: Biological: GamCovidVac vector vaccine for the prevention of COVID-19 (with altered antigenic profile)

INTERVENTIONS:
Biological: GamCovidVac vector vaccine for the prevention of COVID-19 (with altered antigenic profile) — Two intramuscular injections of the GamCovidVac vector vaccine for the prevention of COVID-19 (with altered antigenic profile) will be performed. 1st injection - component I, 2nd injection - component II.

SUMMARY:
Safety, reactogenicity and immunogenicity study of the vector vaccine GamCovidVac for the prevention of coronavirus (COVID-19) infection caused by the SARS-CoV-2 virus with altered antigenic profile with participation of adult volunteers

ELIGIBILITY:
Inclusion Criteria:

The study will include volunteers who meet all the specified criteria:

1. Written informed consents to participate in the Study;
2. Adult volunteers men and women over 18 years old;
3. A negative test result for COVID-19, determined by PCR or express method before the introduction of the investigational medicinal product (IMP);
4. Consent to the use of effective methods of contraception during the entire period of participation in the Study;
5. A negative pregnancy test based on the results of a urine test at a screening visit (for women with preserved reproductive potential);
6. Negative test for the presence of narcotic and psychostimulants in the urine at the screening visit;
7. Negative alcohol content test at the screening visit;
8. Any vaccination not earlier than the last 30 days before inclusion in the Study;
9. No contraindications to vaccination;
10. Absence of acute infectious and/or respiratory diseases for at least 14 days prior to inclusion in the Study.

Exclusion Criteria:

Volunteers cannot be included in the Study if there is at least one of the following criteria for non-inclusion:

1. No written informed consents to participate in the Study
2. Therapy with steroids (with the exception of hormonal contraceptives and/or hormone replacement therapy) and / or immunoglobulins or other blood products that did not end 30 days before inclusion in the Study;
3. Therapy with any immunosuppressive drugs completed less than 3 months prior to inclusion in the Study;
4. Female volunteers during pregnancy or lactation;
5. Acute coronary syndrome or stroke suffered less than one year prior to inclusion in the Study;
6. Tuberculosis, chronic systemic infections (according to anamnesis);
7. Burdened allergic anamnesis (record of anaphylactic shock, Quincke's edema, polymorphic exudative eczema, serum sickness in the anamnesis), hypersensitivity or allergic reactions to the administration of immunobiological drugs, known allergic reactions to any of the components of the vaccine or vaccine containing similar components, exacerbation of allergic diseases on the day of inclusion in the Study;
8. The presence of neoplasms (ICD codes C00-D09) (according to anamnesis);
9. Splenectomy (according to the anamnesis);
10. Neutropenia (decrease in the absolute number of neutrophils less than 1000 cells / mm3), agranulocytosis, significant blood loss, severe anemia (hemoglobin concentration less than 80 g/l) - 6 month prior to inclusion in the Study (according to the anamnesis);
11. Volunteers with an active form of the disease caused by the human immunodeficiency virus, syphilis, hepatitis B and C (according to the anamnesis);
12. Anorexia, protein deficiency of any origin;
13. Alcoholism and drug addiction (according to the anamnesis);
14. Participation in any other clinical trial 90 days prior to the screening;
15. Extensive tattoos at the injection sites (deltoid muscle area), which do not allow to assess the local reaction to the introduction of investigational medicinal product (IMP);
16. Any other condition of the volunteer of the Study, which, in the opinion of the research physician, may prevent the completion of the study in accordance with the protocol;
17. Vaccination against COVID-19 or transmitted coronavirus infection (COVID-19) less than 6 months prior to the screening;
18. Multiple administration of the Sputnik V vaccine, Sputnik Lite, or multiple administration of any other COVID-19 vaccine for more than three injections (Sputnik V vaccination plus Sputnik Lite revaccination);
19. Inability to read in Russian; inability or unwillingness to understand the essence of the Study;
20. Any other conditions that limit the validity of obtaining informed consent or may affect the ability of a volunteer to participate in the Study.
21. Staff of research centers (chief researcher and members of the research team) directly involved in the research and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AE) | Within 28 days after administration of the drug
  Occurrence of adverse events (AE)
Occurrence of serious adverse events (SAEs) | Throughout Study completion, until December 2024
  Occurrence of serious adverse events (SAEs)

IPD SHARING:
Plan to Share IPD: Undecided